CLINICAL TRIAL: NCT05654194
Title: A Single Arm Study to Evaluate the Safety and Efficiency of Azacitidine (AZA) Combination With Venetoclax and ATRA in Patients With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: Azacitidine Combined With Venetoclax and ATRA in Newly Diagnosed AML
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOOCHOW-HY-2022-11-2
Record Dates: First submitted 2022-11-25; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Azacitidine; Venetoclax; ATRA
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AVA（Azacitidine Combined With Venetoclax and ATRA）group (Experimental): (1)Inductive therapy: AZA 75mg/m² per day for days 1-7 and venetoclax 100mg orally for day 2 , 200mg orally for day 3, 300mg orally for day4-6, 400mg orally for day7-10,ATRA 45mg/m² for day 12-28,every 28 days for up to 2 cycles or progression; (2)Consolidate therapy:ATRA 45mg/m2 per day for d1-21 ,AZA 70mg/m² per day for days 1-7, every 28 days for up to 4 cycles or progression; (3) Maintenance therapy:ATRA 45mg/m2 for d1-21 every 28 days,AZA 70mg/m² per day for days 1-7, every 3 month untill progression;
  Interventions: Drug: Azacitidine Combined With Venetoclax and ATRA group

INTERVENTIONS:
Drug: Azacitidine Combined With Venetoclax and ATRA group — AZA 75mg/m² per day for days 1-7 and venetoclax 100mg orally for day 2 , 200mg orally for day 3, 300mg orally for day4-6, 400mg orally for day7-10,ATRA 45mg/m² for day 12-28,every 28 days for up to 2 cycles as the inductive therapy.ATRA 45mg/m2 per day for d1-21 ,AZA 70mg/m² per day for days 1-7, every 28 days for up to 4 cycles for consolidate therapy.ATRA 45mg/m2 for d1-21 every 28 days,AZA 70mg/m² per day for days 1-7, every 3 month for Maintenance therapy
  Other Names: AVA group

SUMMARY:
This is a single arm study to evaluate the safety and efficiency of azacitidine (AZA) combination with venetoclax and ATRA in Patients With Newly diagnosed acute myeloid leukemia. Azacitidine, venetoclax and ATRA, may stop the growth of cancer cells, either by demethylation, by promoting cells differentiation or by killing the cells.

DETAILED DESCRIPTION:
This study include newly diagnosed AML patients who will accept the therapy with AZA combined with venetoclax and ATRA: (1)Inductive therapy: AZA 75mg/m² per day for days 1-7 and venetoclax 100mg orally for day 2 , 200mg orally for day 3, 300mg orally for day4-6, 400mg orally for day7-10,ATRA 45mg/m² for day 12-28, every 28 days for up to 2 cycles or progression; (2)Consolidate therapy:ATRA 45mg/m2 per day for d1-21 ,AZA 70mg/m² per day for days 1-7, every 28 days for up to 4 cycles or progression; (3) Maintenance therapy:ATRA 45mg/m2 for d1-21 every 28 days,AZA 70mg/m² per day for days 1-7, every 3 month till progression;

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML according to the WHO (2016) classification of acute myeloid leukemia.
* Age ≥ 18years.
* ECOG score: 0-3.
* White blood cell count ≤ 25*10^9/L
* Total bilirubin ≤ 3X the institutional upper limit of normal if attributable to hepatic infiltration by neoplastic disease
* AST (SGOT) and ALT (SGPT) ≤ 3X the institutional upper limit of normal
* Creatinine clearance ≥30ml/min

Exclusion Criteria:

* Pregnancy or lactation.
* Acute promylocytic leukemia or chronic myeloid leukemia in blast crisis.
* Another malignant disease.
* Uncontrolled active infection.
* Left ventricular ejection fraction < 0.3 by echocardiography or grade III/IV cardiovascular dysfunction according to the New York Heart Association Classification.
* Active hepatitis B or hepatitis C infection.
* HIV infection.
* Other commodities that the investigators considered not suitable for the enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of the bone marrow complete response | after completion of one induction courses (1st Induction Course is 28 days) and before starting of the 2nd cycle
  Rate of the bone marrow complete response after 1 cycle of inductive therapy include Rate of the bone marrow complete response included the rate of the including Complete Remission(CR) and Complete Remission with incomplete hematologic recovery (CRi) after 1 cycle of inductive therapy

SECONDARY OUTCOMES:
Rate of the bone marrow complete response after 2 cycle of inductive therapy | after completion of two induction courses (1st Induction Course is 28 days) and before starting of the 1st Consolidation cycle
  Rate of the bone marrow complete response after 2 cycle of inductive therapy include Rate of the bone marrow complete response included the rate of the including Complete Remission(CR) and Complete Remission with incomplete hematologic recovery (CRi) after 2 cycle of inductive therapy
Minimal Residual Disease (MRD) response | after completion of two induction courses (one Course is 28 days) and before starting of the 1st Consolidation cycle
  MRD response in bone marrow at the end of 2nd cycle
Overall Survival (OS) | 2 years
  time from randomization to death from any cause
Event Free Survival（EFS） | 2 years
  time from randomization to the relapse ,death or drug is unacceptably toxic
Number of adverse events | 2 years
  adverse events are evaluated with CTCAE V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Han, PhD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- the First Affiliated Hospital of Soochow University, Suzhou, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/94/NCT05654194/ICF_000.pdf